CLINICAL TRIAL: NCT00918541
Title: Natural 1-year History of Atherosclerosis in Asymptomatic Patients With Mild to Moderate Carotid Stenosis
Brief Title: Natural History of Atherosclerosis
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Districthospital of Bellinzona (Unknown)
Responsible Party: Sponsor
Other Study IDs: CarotidMRI
Record Dates: First submitted 2008-11-19; First posted 2009-06-11 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Atherosclerosis
Keywords: atherosclerotic disease; progression; natural progression of atherosclerotic disease; natural history of atherosclerosis at the level of the carotid artery as evaluated by MRI
MeSH Terms: conditions — Atherosclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: asymptomatic patients with mild to moderate carotid artery stenosis

SUMMARY:
20 patients will be recruited. The aim of the study is to determine the natural progression of atherosclerotic disease.

ELIGIBILITY:
Inclusion Criteria:

* stable carotid artery disease not requiring revascularization
* asymptomatic carotid artery stenosis < 80% or symptomatic patients with stenosis < 60 %
* prophylactic therapy with aspirin (> 100mg/day, statin, blood pressure therapy if indicated (goal < 130/80 mmHg))
* informed consent

Exclusion Criteria:

* non atherosclerotic occlusive disease (Bürgers disease)
* uncontrolled BP (DBP > 110 mmHg and/or SBP > 200 mmHg)
* hemorrhagic disease or platelet count < 100'000 mm^3
* Known active liver disease (elevations of GPT GOT or increased ammonia)
* impaired renal function (crea > 180 mmol/l)
* pregnancy
* severe claustrophobic reactions
* short - term life - threatening pathology
* physically unable to participate in the study
* compliance not guaranteed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the districthospital Bellinzona
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Progression of atherosclerotic plaque | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Corti, MD, Principal Investigator — Cardiovascular Center Cardiology, University Hospital Zürich, Zürich Switzerland; Augusto Gallino, MD, Principal Investigator — Ospedale San Giovanni Bellinzona, Switzerland
Locations (3):
- Switzerland (3):
  - Ospedale San Giovanni Bellinzona, Bellinzona
  - Ospedale San Giovanni, Bellinzona
  - Cardiovascular Center Cardiology University Hospital Zürich, Zurich